CLINICAL TRIAL: NCT04925466
Title: Comparison of 10cmH2O and Manual Titrated Pressure in Treatment of Obstructive Sleep Apnea(OSA) Patients
Brief Title: Acceptable Pressure Range for Continuous Positive Airway Pressure(CPAP) Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State Key Laboratory of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Yuan-Ming Luo, Proffessor, State Key Laboratory of Respiratory Disease
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2021016
Record Dates: First submitted 2021-06-04; First posted 2021-06-14 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Obstructive Sleep Apnea of Adult
Keywords: OSA; CPAP; acceptable range

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with CPAP at 10cmH2O (Experimental): Patients with OSA will be treated with CPAP at 10cmH2O during sleep.
  Interventions: Device: CPAP at pressure of 10 cmH2O
- Treatment with CPAP at minimal effective pressure (Experimental): Patients with OSA will be treated with CPAP at minimal effective pressure derived from manual titration during sleep.
  Interventions: Device: CPAP at minimal effective pressure

INTERVENTIONS:
Device: CPAP at pressure of 10 cmH2O — Patients used CPAP with the pressure of 10 cmH2O during overnight polysomnography
  Arms: Treatment with CPAP at 10cmH2O
Device: CPAP at minimal effective pressure — Patients with OSA will be treated with CPAP at minimal effective pressure derived from manual titration during sleep.
  Arms: Treatment with CPAP at minimal effective pressure

SUMMARY:
Compliance of continuous positive airway pressure （CPAP） derived from auto-titration is similar to that derived from manual titration, although pressure derived from the former was usually 2-5 cmH2O higher than the latter. Therefore the Investigators hypothesize that accurate titration maybe not necessary for successful treatment of obstructive sleep apnea (OSA) as long as CPAP pressure was not lower than the minimal effective pressure.

DETAILED DESCRIPTION:
Study Design: A randomized, cross-over and double-blind study. Objective: To compare the pressure of 10 cmH2O and minimal effective pressure derived from manual titration on the effect of CPAP treatment in OSA. Methods: Patients with suspected OSA (age, body mass index and symptom) to be referred to a sleep centre were recruited. Patients with OSA confirmed by overnight full polysomnography (PSG) were invited to do standard overnight manual titration under PSG based on the Academy of Sleep Medicine (AASM) manual guidelines. Patients whose manual titration pressure lower than 10cmH2O and willing to participate in the study were invited to repeat two more nights (3th PSG and 4th PSG) under CPAP pressure at both 10cmH2O and the pressure derived from manual titration in random order. The sleep apnea-hypopnea index (AHI), obstructive sleep apnea index (OHI), arousal index (ArI), oxygen desaturation index (ODI), sleep structure, and treatment preference were to be observed.

ELIGIBILITY:
Inclusion Criteria:

1. reported snore, apnea and daytime sleepiness;
2. a diagnosis of obstructive sleep apnea with polysomnography according to ASSM guideline(apnoea-hypopnea-index(AHI)≥5 events/h) and need to be treated with continuous positive airway pressure;
3. willing to participate after informed consent.

Exclusion Criteria:

1. Evidence of severe coronary or cerebral, cardiovascular disease and significant memory, perceptual or behavioural disorder;
2. Severe respiratory disease defined as severe chronic obstructive pulmonary disease(ie. FEV1/FVC<70% and FEV1<50%predicted) or resting awake SaO2<90%
3. Have known contraindications with CPAP, like current pneumothorax and hemoptysis, et al.
4. Central sleep apnea>10 events/h；
5. Frequent nasal congestion；
6. Optimal treatment CPAP pressure(by manual titration) equal or higher than 10cmH2O.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-05 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
sleep structure | 4 full night
  Assessment of the sleep efficiency (percentage is calculated by dividing Total Sleep Time by Total Time in bed)
arousal index | 4 full night
  total number of arousal events/total sleep time(h)
Apnea hypopnea index | 4 full night
  Total number of apneas and hypopneas/total sleep time (h)
Oxygen Desaturation Index | 4 full night
  Total number of oxygen desaturations≥3% /total sleep time(h)

SECONDARY OUTCOMES:
Patients preference | 4 full night
  Using a questionnaire named preference to record patients preference to 10cmH2O or manual titrated pressure

CONTACTS AND LOCATIONS:
Overall Officials: Yuanming Luo, PhD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang L, Chen Y, Wei Q, Wu Y, Huang C, Liang S, Steier J, Catcheside P, Eckert D, Wellman A, Luo Y. Fixed CPAP at 10 cmH 2O May Replace Manual Titration in Moderate to Severe OSA Patients: A Preliminary Randomised Controlled Trial. Respirology. 2025 Aug;30(8):770-778. doi: 10.1111/resp.70037. Epub 2025 Mar 25. PMID 40130675